CLINICAL TRIAL: NCT06670794
Title: Using Ecological Momentary Data to Inform a Web Intervention for Romantic Partners Concerned About Their Loved Ones' Drinking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Stanford University (Other); Portland State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202401222; 1R34AA030182-01A1 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-06-30 (Actual); Status verified 2025-06

CONDITIONS: Experimental; Control Condition
Keywords: alcohol; alcohol use disorder; community reinforcement and family training; concerned partners; concerned significant others; communication
MeSH Terms: conditions — Alcoholism; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation control (Other): Psychoeducation control CPs will be routed to visit self-help resources on NIAAA's website ("Alcohol's Effects on Health") and asked to spend the same amount of time (20-30 minutes) reviewing site content.
  Interventions: Behavioral: Psychoeducation control
- Experimental web-based intervention (Experimental): CPs in the experimental web-based intervention condition will complete web-based sessions including personalized feedback and information about how communication and self-care affect their own well-being and their partner's alcohol use behaviors.
  Interventions: Behavioral: Web-based intervention for concerned partners

INTERVENTIONS:
Behavioral: Web-based intervention for concerned partners — The web-based intervention will comprise sessions focusing on community reinforcement and family therapy principles including: (1) self-care, (2) positive communication including ways to increase responsiveness to their partner (PPR; i.e., actively listening, showing understanding, expressing interest in what their partner is thinking and feeling, and trying to see where their partner is coming from), (3) understanding their partner's drinking reinforcers, and (4) supporting their partner if they want help and engaging in positive, healthy activities with their partner.
  Arms: Experimental web-based intervention
Behavioral: Psychoeducation control — This is a psychoeducation control condition.
  Arms: Psychoeducation control

SUMMARY:
Aim 1. Couples (N=50 dyads) with a Concerned Partner (CP) and a Drinking Partner (DP) will independently complete baseline and follow-up surveys and a 21-day EMA with three daily reports on their communication and DP's drinking. Aim 2. Iteratively develop a four-session web based intervention and evaluate the WBI's feasibility and acceptability with 15 CPs. Aim 3. Perform a pilot randomized controlled trial (RCT) comparing WBI to psychoeducation control in 110 couples.

DETAILED DESCRIPTION:
Alcohol misuse negatively affects relationships and is significantly correlated with higher rates of relationship conflict, distress, and dissolution as well as other serious negative interpersonal consequences (e.g., domestic violence, sexual assaults). Encouragement from concerned partners (CPs) is a common motivator for those who misuse alcohol to pursue care and often the most helpful mechanism in supporting change. The goals of this proposal are to: Identify how specific CP behaviors influence their partner's alcohol craving, motives, drinking, and problems on a daily basis using dyadic ecological momentary assessment techniques (Aim 1); use the knowledge from EMA analysis to iteratively develop a CP-focused web-based intervention (WBI) that provides psychoeducation about communication patterns that influence DP drinking and by integrating personalized feedback about CPs' own communication behaviors that may be working against their goals (Aim 2); and pilot the WBI's efficacy on CP outcomes (depression, anxiety, social support), their partner's drinking behavior (alcohol consumption, motives, related consequences), and both partners' relationship distress and conflict (Aim 3). The investigators expect the WBI will yield significant improvements in all outcomes. This project is significant because intervening with CPs has strong potential to change relationship dynamics that may reduce problems and prevent future problems associated with alcohol misuse. It also develops a new prevention model that does not rely on the drinking partner attending a clinical facility to access care. The proposed study is innovative because it uses dyadic and ecological momentary assessment designs to test dynamic questions about interdependence in relationship interactions and alcohol use between partners and employs the generated knowledge to inform intervention adaptation. Teaching CPs to effectively communicate their concerns may be a necessary catalyst for decreasing their partner's alcohol use and preventing alcohol use disorders. The potential reach of this intervention is large such that it can be easily implemented over the web to those who may need help but would not otherwise seek care.

ELIGIBILITY:
CP Inclusion Criteria:

* be at least 18 years old
* be in a romantic relationship with their partner
* be living with their partner,
* have a computer, tablet, or mobile phone with Internet access
* have no plans to separate from their partner in the next 60 days
* indicate no concerns they would be physically hurt by their partner on the Intimate Partner Screen

CP Exclusion Criteria:

* drinking scores at or above the threshold for DP participation

DP Inclusion Criteria:

* be at least 18 years old
* misuses alcohol as defined by their scores (4+ for women/non-gender confirming, 5+ for men) on the consumption portion of the Alcohol Use Disorder Identification Test (AUDIT-C) (Dawson et al., 2005)
* has a computer, tablet, or mobile phone with Internet access
* indicates no concerns they would be physically hurt by their partner

DP Exclusion Criteria:

* current alcohol treatment
* currently concerned about their partner's drinking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CP Depression Symptoms Questionnaire | 1 month post-intervention.
  Patient Health Questionnaire. 8 items. Scores range from 0-32. Higher scores indicate more depressive symptoms.
CP Anxiety Symptoms Questionnaire | 1 month post-intervention.
  Generalized Anxiety Disorder scale. 7 items. Higher scores indicate more anxiety symptoms.
CP Anger expression questionnaire | 1 month post-intervention.
  Dimensions of Anger Reactions - 5 item (DAR-5). Scores range 1-5 with higher scores indicating greater anger.
CP Loneliness Questionnaire | 1 month post-intervention.
  Measure: UCLA 3-item Loneliness Scale (Hughes, M. E., Waite, L. J., Hawkley, L. C., & Cacioppo, J. T. (2004). A Short Scale for Measuring Loneliness in Large Surveys. Research on Aging, 26(6), 655-672. https://doi.org/10.1177/0164027504268574) Scores are 1-9. Higher scores indicate more loneliness.
CP Partner Social Support Questionnaire | 1 month post-intervention.
  Marital Perceived Social Support (Cohen et al., 1985). Scored 0-3. Higher scores mean more social support.
CP-DP Relationship Functioning Questionnaire | 1 month post-intervention.
  Quality of Marriage Index (Norton, 1983). Higher scores indicate greater relationship satisfaction.
DP AUDIT Questionnaire | 1 month post-intervention.
  Drinking Partner's AUDIT score. 10 items. Items are summed. Greater scores indicate greater alcohol use.
CP General Social Support Questionnaire | 1 month post-intervention.
  MOS Social Support Survey (Sherbourne & Stewart, 1991). Scored 1-5. Higher scores indicate more social support. Sherbourne, C. D., & Stewart, A. L. (1991). The MOS social support survey. Social science & medicine, 32(6), 705-714.
DP Alcohol Use Questionnaire | 1 month post-intervention.
  Drinking Partner's:
  Alcohol consumption via the Quantity/Frequency/Peak Alcohol Use Index (Dimeff et al., 1991). Six items measure the drinking partner's alcohol consumption. The items are not scored together but evaluated individually (e.g., frequency, typical quantity, peak quantity, etc.). Higher scores denote greater consumption.
DP Drinking Motives Questionnaire | 1 month post-intervention.
  Drinking Partner's Drinking Motives using the Drinking Motives Questionnaire (Cooper et al., 1992). Subscales for coping, enhancement, social, and conformity. Items are averaged. Higher scores indicate greater endorsement of that motive.
DP Alcohol-related Consequences Questionnaire | 1 month post-intervention.
  Drinking Partner's Alcohol-related Consequences assess via the Brief Young Adult Alcohol Related Consequences measure. 24 items. Scores are created by summing the items. Higher scores denote greater consequences endorsed.

SECONDARY OUTCOMES:
CP-DP Communication Questionnaire | 1 month post-intervention.
  Family Environment via the Brief Family Relationship Scale. Fok, C. C., Allen, J., Henry, D., & People Awakening Team (2014). The brief family relationship scale: a brief measure of the relationship dimension in family functioning. Assessment, 21(1), 67-72. https://doi.org/10.1177/1073191111425856. Cohesion, expressiveness, and conflict subscales. Items are averaged. For each subscale, greater scores reflect greater cohesion, expressiveness, and constructive ways of handling conflict.
CP-DP Perceived Partner Responsiveness Questionnaire | 1 month post-intervention.
  Measures perceived partner responsiveness. Scores range from 1-5. Greater scores mean greater responsiveness perceived about the partner.
  Source articles:
  Laurenceau, J. P., Barrett, L. F., & Pietromonaco, P. R. (1998). Intimacy as an interpersonal process: The importance of self-disclosure, partner disclosure, and perceived partner responsiveness in interpersonal exchanges. Journal of Personality and Social Psychology, 74(5), 1238-1251. https://doi.org/10.1037//0022-3514.74.5.1238 O'Neill, A.S., Mohr, C.D., Bodner, T., & Hammer, L. (2020). Perceived Partner Responsiveness, Sleep and Pain: A Dyadic Study of Military-Connected Couples. Health Psychology, 39(12), 1089-1099. https://doi.org/10.1037/hea0001035
CP Communication about Drinking Questionnaire | 1 month post-intervention.
  We have created a measure adapted from the Spouse Behavior Questionnaire (Love et al., 1991) and the Partner Management Strategies Questionnaire (Rodriguez et al., 2013) that will assess different behaviors CPs use to attempt to change their partner's drinking. Subscales include punishing drinking, rewarding sobriety, withdrawing, and supporting drinking. Items are averaged. Higher scores mean greater endorsement of these subscales.
CP-DP Communication: Number of conflicts | 1 month post-intervention.
  We will ask participants the number of disagreements they have had with their partner. Higher numbers denote more disagreements.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Rodriguez, Ph.D., Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: Yes
The data will be deidentified, but shared data will be at the individual level.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 2 years of the award end date, as required by the NIAAA Data Archive. Data will also be grouped based on publication, which will be shared when the pre-print is available. These publications will have DOIs to aid in findability. Raw data will include a GUID to help with indexing. The NIAAA Data Archive will make decisions about how long to preserve data.
Access Criteria: Any scientific researcher may access our de-identified data, as consistent with the NIAAA Data Archive. To request access of the data, researchers will use the standard processes for the NIAAA Data Archive, and the Data Access Committee will decide which requests to grant. The standard NIAAA data access process allows access for one year and is renewable. Data will be findable for the research community through utilization of the NIAAA Data Archive, which is a public data repository housed under the NIMH. All participants will be assigned a GUID to allow for standard indexing. Research publications and manuscripts will be assigned a digital object identifier (DOI), which will be referenced in the data, to allow for the research community to access the exact information used for this publication.